CLINICAL TRIAL: NCT05669183
Title: Comparison of Peripheral and Central Intubation on Hemodynamics in Veno-arterial-extracorporeal Membrane Oxygenation (RECOVERY): a National, Multi-center, Prospective, Cohort Study
Brief Title: Hemodynamic Comparison of Peripheral and Central VA ECMO.
Acronym: RECOVERY
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Peking University Third Hospital (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Beijing Anzhen Hospital (Other); Guangdong Provincial People's Hospital (Other); Shaanxi Provincial Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2021CRF-005
Record Dates: First submitted 2022-10-30; First posted 2022-12-30 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Shock, Cardiogenic; Cardiac Arrest; Extracorporeal Circulation; Complications; Hemodynamics Instability
MeSH Terms: conditions — Shock, Cardiogenic; Heart Arrest | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Peripheral VA ECMO: Femoral artery cannulation for veno-arterial extracorporeal membraneous oxygenation (VA ECMO)
  Interventions: Procedure: Veno-arterial extracorporeal membrane oxygenation
- Central VA ECMO: Axillary artery cannulation for veno-arterial extracorporeal membraneous oxygenation (VA ECMO)
  Interventions: Procedure: Veno-arterial extracorporeal membrane oxygenation

INTERVENTIONS:
Procedure: Veno-arterial extracorporeal membrane oxygenation — Veno-arterial extracorporeal membrane oxygenation (VA ECMO) is mainly used for circulatory support in patients with severe cardiopulmonary failure. VA ECMO drains the blood from the venous system followed pumping the blood back into the arterial vascular compartment after oxygenation. It can be divided into two cannulation strategies for VA ECMO support, namely peripheral VA ECMO and central VA ECMO based on the arterial cannulation site. Peripheral VA ECMO is established via the femoral artery (FA), whereas axillary artery (AX) is an arterial cannulation site in central VA-ECMO.

SUMMARY:
The goal of this clinical trial is to monitor hemodynamic differences between central veno-arterial extracorporeal membrane oxygenation (VA ECMO) and peripheral VA ECMO. The main question it aims to answer is:

* Efficacy of the different cannulation strategies for the establishment of for VA-ECMO circulation on hemodynamics and organ perfusion.

Participants require VA ECMO support, will be divided into two groups in an intention-to-treat analysis: central artery cannulation and peripheral artery cannulation.

Researchers will analyze different cannulation strategies for VA-ECMO and identify potential advantages and disadvantages for two groups of VA-ECMO.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years
* Participants with cardiogenic shock
* Obtaining informed consent from participants or their affiliated beneficiaries

Exclusion Criteria:

* Irreversible heart failure
* Contraindications to anticoagulation therapy
* Uncontrolled bleeding
* Irreversible neurological pathology
* Participants limited to extracorporeal cardiopulmonary resuscitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants require VA ECMO support for cardiogenic shock or cardiac arrest.
Sampling Method: Probability Sample
Enrollment: 136 (Estimated)
Dates: Start 2023-08-12 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Oxygen saturation-no. (%) | Through VA ECMO support completion, an average of 1 week
  Blood gas analysis
Left ventricular end-diastolic volume (ml) | Through VA ECMO support completion, an average of 1 week
  echocardiography
Left ventricular End-systolic volume (ml) | Through VA ECMO support completion, an average of 1 week
  echocardiography
Stroke volume (ml) | Through VA ECMO support completion, an average of 1 week
  echocardiography
Mitral valve area(cm2) | Through VA ECMO support completion, an average of 1 week
  echocardiography

SECONDARY OUTCOMES:
Rate of successful weaning from VA ECMO | Through study completion, up to 2 years
  Weaning success is defined as survival after complete removal of the extracorporeal circuit without requirement for further mechanical support or heart transplant.
VA ECMO duration | Through VA ECMO support, an average of 1 week
  Length of VA ECMO support
Cannulation-related complications | Through study completion, up to 2 years
  Cannulation-related complications include bleeding, limb ischemia, revision of cannulation site, wound complications. Limb ischemia is defined as ischemia requiring any surgical procedure, including revision of the arterial/distal perfusion cannula, fasciotomy for compartment syndrome, gangrene, or amputation. Wound complication is defined as infection or requirement of an additional surgical intervention, such as arterial repair, washout with or without vacuum-assisted closure, and muscle flap closure.
Duration of ICU stay | Through study completion, up to 2 years
  Intensive care unit length of stay
Duration of hospital stay | Through study completion, up to 2 years
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yan, Study Director — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No